CLINICAL TRIAL: NCT06824415
Title: Optimizing Depression Treatment Through Sleep-state Brain Stimulation
Brief Title: Sleep TMS for Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Corey Keller, Associate Professor in Department of Psychiatry and Behavioral Sciences, Stanford University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 60980-3; UM1TR004921 (NIH)
Record Dates: First submitted 2025-02-07; First posted 2025-02-13 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Major Depression; Sleep
Keywords: sleep; tms; eeg
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active TMS, Sham TMS (Experimental): Participants will receive 2 sessions of Transcranial Magnetic Stimulation (TMS) delivered using standard intermittent theta-burst (iTBS) parameters (600 pulses, 3 min, 120% rMT). Participants will receive, on separate sessions, either active or sham iTBS delivered during pre-sleep wakefulness or NREM sleep stages while recording with Electroencephalography (EEG). Participants will perform the N-back task and Multi-source Interference Task (MSIT) during each session to measure working memory and cognitive control performance.
  Interventions: Device: TMS
- Sham TMS, Active TMS (Experimental): Participants will receive 2 sessions of Transcranial Magnetic Stimulation (TMS) delivered during using standard intermittent theta-burst (iTBS) parameters (600 pulses, 3 min, 120% rMT). Participants will receive, on separate sessions, either active or sham iTBS delivered during pre-sleep wakefulness or NREM sleep stages while recording with Electroencephalography (EEG). Participants will perform the N-back task and Multi-source Interference Task (MSIT) during each session to measure working memory and cognitive control performance.
  Interventions: Device: TMS

INTERVENTIONS:
Device: TMS — Transcranial magnetic stimulation (TMS) applies magnetic pulses to stimulate nerve cells in the brain.

SUMMARY:
The goal of this study is to establish the feasibility, tolerability, and preliminary efficacy of sleep-state transcranial magnetic stimulation (TMS) for enhancing plasticity in depression treatment.

ELIGIBILITY:
Inclusion Criteria:

* Current Major Depressive Disorder (MDD) diagnosis
* Failed >= 1 antidepressant medication
* Moderate-to-severe depression

Exclusion Criteria:

* Intellectual disability
* Significant head injury/neurological disorder
* Pregnancy or postpartum
* TMS/MRI contraindications
* Active substance use/suicidal ideation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Baseline TMS-EEG after iTBS | Baseline, end of iTBS (3 minutes)
  Changes in Early Local TMS-Evoked Potentials (EL-TEP) following 3 minutes of either active or sham iTBS in each session to assess cortical excitability and plasticity measures.
  1) tbs; 2) sleep (cortical excitability and plasticity measures) in both active and sham.
Change in Baseline TMS-EEG after NREM Sleep | Baseline, end of sleep stage (3 hours)
  Changes in Early Local TMS-Evoked Potentials (EL-TEP) following 3 hours of NREM sleep in each session to assess cortical excitability and plasticity measures.
Change in N-back Accuracy Performance | Baseline, end of sleep stage (3 hours)
  N-back task (15-min) measures working memory performance and accuracy will be determined by the number of correct responses to the stimulus. Change in accuracy performance will be assessed before and after NREM sleep.
Change in N-back Reaction Time Performance | Baseline, end of sleep stage (3 hours)
  N-back task (15-min) measures working memory performance and reaction time will be determined by the time it takes for the participant to respond to the stimulus. Change in reaction time performance will be assessed before and after NREM sleep.
Change in MSIT Accuracy Performance | Baseline, end of sleep stage (3 hours)
  Multi-source Interference Task (MSIT; 15-min) measures cognitive control performance and accuracy will be determined by the number of correct responses to the stimulus. Change in accuracy performance will be assessed before and after NREM sleep.
Change in MSIT Reaction Time Performance | Baseline, end of sleep stage (3 hours)
  Multi-source Interference Task (MSIT; 15-min) measures cognitive control performance and reaction time will be determined by the time it takes for the participant to respond to the stimulus. Change in reaction time performance will be assessed before and after NREM sleep.

SECONDARY OUTCOMES:
Changes in Pittsburgh Sleep Quality Index (PSQI) Scores | After each sleep session (3 hours)
  The Pittsburgh Sleep Quality Index (PSQI) contains 19 self-rated questions which measures seven aspects of sleep: (1) subjective sleep quality, (2) sleep latency, (3) sleep duration, (4) habitual sleep efficiency, (5) sleep disturbances, (6) use of sleeping medication, and (7) daytime dysfunction. The 19 self-rated items are combined to form seven component scores, each of which has a range of 0-3 points (0 indicates no difficulty, while 3 indicates severe difficulty). The seven component scores are then summed to yield one global score, with a range of 0-21 points (0 indicating no difficulty, and 21 indicating severe difficulties in all the seven areas of sleep quality).
Changes in Treatment Tolerability | After each sleep session (3 hours)
  Treatment tolerability will be assessed through subject-reported comfort ratings on loudness, scalp sensation, and pain perception on scales ranging from 0 to 10.

CONTACTS AND LOCATIONS:
Overall Officials: Corey J Keller, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No